CLINICAL TRIAL: NCT01978379
Title: The Nociception Level During Anesthesia in Patients Undergoing Video-assisted Thoracoscopic Surgery
Brief Title: The Nociception Level During General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Srdjan Jelacic, Acting Assistant Professor, University of Washington
Other Study IDs: 44750-B
Record Dates: First submitted 2013-10-25; First posted 2013-11-07 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Pain
Keywords: General Anesthesia; Nociception Level
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We are conducting a study to evaluate two investigational devices that may help us better monitor discomfort or pain in anesthetized patients during minimally invasive lung surgery. We want to collect information on how people respond to pain related to their surgery. Currently, we use blood pressure (BP) and heart rate (HR) to check the response to pain. In this study, we will also use two devices called the Medasense PMD-100 and PhysioDoloris monitors to look at measurements of pain. We will compare the measurements from the study devices to the measurements of heart rate and blood pressure. We hope to enroll about 40 subjects in this study at the University of Washington Medical Center.

DETAILED DESCRIPTION:
The following measurements will be collected during surgery for this research study.

1. Nociception Level (NoL) index The PMD-100 monitor includes a small probe similar to the pulse oximeter that will be placed on the subjects finger, which will be connected to the laptop placed next to the anesthesia machine. We will measure and record NoL index values at the following painful events: placement of breathing tube, skin incision, initial surgical instruments insertion and muscle relaxation assessment with a twitch monitor (60mA, 100Hz, 30sec). The anesthesiologist will be blinded to NoL index values that will only be collected for research purposes. We will compare the NoL index to ANI index, BP and HR. The measurements will start 5 minutes prior to the administration of general anesthesia and will continue until 5 min. after initial surgical instruments insertion.
2. Analgesia Nociception Index (ANI) index The PhysioDoloris monitor attached to the IV pole will be connected with a cable to the anesthesia monitor. We will measure and record ANI index values at the following painful events: placement of breathing tube, skin incision, initial surgical instruments insertion and muscle relaxation assessment with a twitch monitor (60mA, 100Hz, 30sec). The anesthesiologist will be blinded to ANI index values that will only be collected for research purposes. The measurements will start 5 minutes prior to the administration of general anesthesia and will continue until 5 min. after initial surgical instruments insertion.
3. Blood Pressure and Heart Rate We will also collect blood pressure and heart rate measurements that are generated as part of the standard anesthesia monitoring from electronic anesthesia record at 30 second intervals.
4. Bispectral Index We will also collect Bispectral Index (BIS) measurements that are generated as part of the anesthesia monitoring from electronic anesthesia record at 30 second intervals. BIS is a monitor of the depth of anesthesia that uses a sensor placed on patient's forehead. BIS monitor calculates a dimensionless number estimating the patient's level of consciousness. The BIS values range from 0 (no brain activity) to 100 (fully awake) with the target range between 40 and 60 for general anesthesia.
5. Pain Medication Data: We will collect the amount of pain medications used during the surgery from electronic anesthesia record.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who clinically consent to elective VATS procedure under general anesthesia,
2. Ages between 18 and 80 years,
3. Able to provide informed consent,
4. English speaking

Exclusion criteria:

1. violation of protocol (e.g., administration of medication that does not comply with the study protocol or inability to measure NoL or ANI index)
2. subject has change of mind
3. surgery has to be repeated.

Non-inclusion criteria:

1. subject refusal
2. non-English speaking
3. previous chronic or neuropathic pain
4. previous chronic use of opioids
5. history of psychiatric disorder
6. previous ipsilateral thoracotomy or VATS
7. morbidly obese with body mass index > 40
8. chronically treated with beta-blockers
9. unable to provide informed consent (we will not enroll subjects that require LAR consent)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective Video-Assisted Thoracoscopic Surgery at University of Washington Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Nociception Level (NoL) index | 5 minutes prior to intubation until 5 minutes after the incision for patients undergoing minimally invasive lung surgery under general anesthesia
  The primary objective of this study is to measure the NoL index in patients having minimally invasive lung surgery and compare it to Analgesia Nociception index (ANI), HR and BP as indicators of pain

SECONDARY OUTCOMES:
Analgesia nociception index (ANI) | 5 minutes prior to intubation until 5 minutes after the incision for patients undergoing minimally invasive lung surgery under general anesthesia
  The secondary objective of this study is to measure the ANI in patients having minimally invasive lung surgery and compare it to NoL index, HR and BP as indicators of pain

CONTACTS AND LOCATIONS:
Overall Officials: Srdjan Jelacic, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Ben-Israel N, Kliger M, Zuckerman G, Katz Y, Edry R. Monitoring the nociception level: a multi-parameter approach. J Clin Monit Comput. 2013 Dec;27(6):659-68. doi: 10.1007/s10877-013-9487-9. Epub 2013 Jul 9. PMID 23835792
- [Background] Logier R, Jeanne M, De Jonckheere J, Dassonneville A, Delecroix M, Tavernier B. PhysioDoloris: a monitoring device for analgesia / nociception balance evaluation using heart rate variability analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:1194-7. doi: 10.1109/IEMBS.2010.5625971. PMID 21095676
- [Derived] Bollag L, Jelacic S, Delgado Upegui C, Wu C, Richebe P. The nociception level index (NOL) response to intubation and incision in patients undergoing video-assisted thoracoscopic surgery (VATS) with and without thoracic epidural analgesia. A pilot study. F1000Res. 2018 Jun 22;7:875. doi: 10.12688/f1000research.15279.1. eCollection 2018. PMID 30026938